CLINICAL TRIAL: NCT02152267
Title: ANALGESIC EFFECT OF CATHODAL TRANSCRANIAL CURRENT STIMULATION OVER RIGHT DORSOLATERAL PREFRONTAL CORTEX IN SUBJECTS WITH MUSCULAR TEMPOROMANDIBULAR DISORDERS: A Double Blind Crossover Randomized Clinical Trial
Brief Title: Analgesic Effect of Cathodal tDCS Over Right DLPFC in Subjects With Muscular TMD: a Double Blind Crossover RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Bahia (Other)
Responsible Party: Principal Investigator, Eduardo Pondé de Sena, Associate Professor of Pharmacology Institute of Health Sciences Federal University of Bahia and Permanent Professor at Postgraduate Program in Interactive Processes of Organs and Systems of the Health and Science Institute of Federal University of Bahia, Federal University of Bahia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 29515714.6.0000.5543
Record Dates: First submitted 2014-05-24; First posted 2014-06-02 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Craniomandibular Disorders
Keywords: Temporomandibular; Musculoskeletal Diseases; Electrical Stimulation of the Brain; Prefrontal Cortex
MeSH Terms: conditions — Craniomandibular Disorders; Musculoskeletal Diseases | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- tDCS 1mA (Experimental): the parameters used in the TDCS will be 1mA, cathodal over right DLPFC and anodal over supraorbital contralateral area.
  Interventions: Device: tDCS
- tDCS 2mA (Experimental): the parameters used in the TDCS will be 2mA, cathodal over right DLPFC and anodal over supraorbital contralateral area.
  Interventions: Device: tDCS
- tDCS Sham (Sham Comparator): the parameters used in the TDCS will be sham, cathodal over right DLPFC and anodal over supraorbital contralateral area.
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — The transcranial direct current stimulation allows the neuronal membranes to neuromodulate and it can enhance or inhibit the potential actions on the cortex. Studies with animals has shown that anodal stimulation modulate the membrane in the way to depolarize which results in a long term potential in the stimulated area
  Other Names: Soterix Medical 1×1 tDCS 1300A

SUMMARY:
1. BACKGROUND: Temporomandibular Disorders (TMD) have become part of the daily routine of all the health care professionals. Some studies have shown improvement in subjects with chronic pain using neuromodulation. Chronic pain is involved with neuronal excitability and the excitatory modulation is also being studied to treat chronic pain. Transcranial direct current stimulation (tDCS) allows the neuronal membranes to be neuromodulated. tDCS can enhance or inhibit the potential actions on the cortex. Studies with animals has shown that anodal stimulation modulate the membrane in the way to depolarize which results in a long term potential in the stimulated area.
2. PROBLEM: Most strategies for the treatment of TMDs are local and aim to treat directly the cranial-facial muscles, applying kinesitherapy on Temporomandibular joint (TMJ) and/or on the jaws and on the occlusion of teeth. Some drugs, such as tricyclic antidepressants, that act in the CNS are used in these patients with positive results in the beginning of the treatment. However, many patients after using these drugs in a daily basis, are refractory to them and do not present an improvement in the pain anymore or present several side-effects. Therefore, the investigators want to know if tDCS over dorsolateral prefrontal cortex (DLPFC) would have an analgesic effect when reaching emotional areas.
3. HYPOTHESIS: The investigators believe that neuromodulation by tDCS over DLPFC would decrease the anxiety level and consequently the muscular hyperactivity that is an important etiological factor of TMD. For that, the masseter motor evoked potential (MEP) will be used to verify any change.
4. AIM: To investigate if cathodal tDCS over right DLPFC has analgesic effects in subjects with muscular TMD.
5. METHOD: The investigators will run a three-arm crossover double blind with 15 muscular TMD subjects. The group treatments will be cathodal tDCS 1mA, cathodal tDCS 2mA and Placebo. To verify selection criteria the investigators will use RDC/TMD, Visual analogical scale (VAS) score from 4 to 10 for six months or longer, Inventory of state-trit anxiety (ISTA) score more than 42. The outcomes will be VAS, sensory testing, Electroencephalogram (EEG) and ISTA.

DETAILED DESCRIPTION:
1. INTRODUCTION Pain is among the main complaints of most patients that seek care in a hospital or a primary care unit. Temporomandibular Disorders (TMD) patients have become part of the daily routine of all the health care professionals. Temporomandibular and cranial-facial disorders are so prevalent that, since 1987, the International Headache Society holds meetings to classify different types of pain associated with head. This resulted in the publication of the Manual of Classification of Headaches - The International Classification of Disorders Headache was revised in 2013.

   There are different strategies to treat TMD patients, and the best is chosen depending on the type of problem diagnosed or the most suitable strategy according to professional experience. Strategies range from advice on lifestyle, psychotherapy, containment of the jaw, kinesitherapy, ultrasound, TENS, muscle relaxants plates, allopathic and homeopathic therapies and surgical interventions to the temporomandibular joint (TMJ). Some of these techniques aim to treat the muscles, others treat the dental occlusion or joint structures and there are those whose primary focus is the psycho-emotional factors. As The TMDs are due to various factors of muscular, joint, emotional, inflammatory, autoimmune or even infectious reasons, the treatment should include different therapies during the rehabilitation process, considering the best strategies for each patient. Literature has shown that the causes of muscular origin are more prevalent in patients with this type of disorder). A systematic review using studies with functional brain imaging, showed that, although the majority of disorders are associated with muscle pain, this would be secondary to a process triggered by the Central Nervous System (CNS). Following this theory, some behavioral studies have shown that the TMD, almost always, are related to preexisting psychopathology.

   Chronic pain is involved with neuronal excitability. a study using transcranial magnetic stimulation (TMS) found higher threshold in both sides of resting motor cortex with lower up regulation responses. Furthermore they found lower responses in the intracortical facilitation and inhibition.

   The transcranial direct current stimulation (tDCS) allows the neuronal membranes to neuromodulate and it can enhance or inhibit the potential actions on the cortex. Studies with animals has shown that anodal stimulation modulate the membrane in the way to depolarize which results in a long term potential in the stimulated area. Some studies have shown improvement in subjects with fibromyalgia and chronic pain using neuromodulation . Some authors suggest anodal tDCS over motor cortex to decrease pain while modulating the activity in the neuronal networks responsible for pain, an example of that is the thalamus. It also facilitates the descending inhibition of pain. However few evidences support the efficacy of tDCS.

   Another montage is tDCS over dorsolateral prefrontal cortex (DLPFC). This area is involved with anxiety and depression without direct analgesic effect. A study showed a pain level decrease after tDCS over DLPFC in patients with emotional and affective troubles. The authors suggested it based on emotional modulation by pain independent networks by somatosensory pain perception. A study found anxiety modulation after tDCS application over DLPFC using cathodal current on the right side and anodal on the left side. This result is just a weak evidence that the tDCS anxiety effect, there is a demand to investigate that approach.

   Regarding the parameters the authors have suggested, 1 or 2mA, but the most common and more used is 2 mA. There is a discussion about which milliamperage is more appropriate when the investigators use cathodal current. A study verified the same results after cathodal and anodal 2mA, both increased the motor evocated potential (MEP) whereas 1mA cathodal current decreased the cortical excitability. Regarding the risks of side and adverse effects a systematic review found just a few adverse effects such as itching, tingling and mild headache that lingered after the stimuli was removed. The adverse effects depend on the intensity and duration and usually the protocol recommends the use of lower intensity (1 or 2mA) during short period of time of 20 or 30 minutes. A questionnaire has been utilized to access these effects.
2. PROBLEM Most strategies for the treatment of TMDs are local and aim to treat directly the cranial-facial muscles, applying kinesitherapy on TMJ and/or on the jaws and on the occlusion. Some drugs, such as tricyclic antidepressants, that act in the CNS are used in these patients with positive results in the beginning of the treatment. However, many patients, after using these drugs in a daily basis, are refractory to them and do not present an improvement in the pain anymore or present several side effects. Therefore, the investigators want to know if tDCS over DLPFC would have an analgesic effect when reaching emotional areas and if there are different results with different amplitude.
3. HYPOTHESIS The investigators believe that neuromodulation by tDCS over DLPFC would decrease the anxiety level and consequently the muscular hyperactivity that is an important etiological factor of TMD. Using the motor evoked potential the investigators will verify if changes will occur after 1mA and 2mA stimulation and if those changes will be different when compared.
4. OBJECTIVES 4.1- GENERAL PURPOSE Investigate if cathodal tDCS over right DLPFC has analgesic effects in subjects with muscular TMD.

   4.2- SPECIFICS PURPOSES 1- Evaluate the tDCS effect regarding pain perception and pressure threshold; 2- Evaluate if tDCS has any effect on anxiety and stress; 3- Measure the masseter MEP pre and post tDCS; 4- Correlate pain intensity with anxiety and masseter MEP pre and post tDCS; 5- Compare tDCS effects over pain intensity, anxiety, stress and masseter MEP after apply different intensities (1mA/2mA).
5. BACKGROUND tDCS has shown promising results for the treatment of chronic pain in several types of diseases, being a good and non-invasive alternative to treat pain in TMD patients. Also, based on studies that showed changes in the brain activity of chronic pain patients and on the difficulties faced to treat TMD, there is a need to conduct clinical trials using new techniques, such as neuromodulation, to help these patients to control their pain. Therefore, tDCS emerges as a new tool to be coupled with other effective treatments already used for these patients. Furthermore, the investigators think that there is a tie relationship between anxiety and muscular hyperactivity but there is no evidence to say that tDCS over emotional areas can decrease anxiety.
6. MATERIALS AND METHODS 6.1 Sample The IMMPACT (Initiative on Methods, Measurement, and Pain Assessment in Clinical Trial) advises an effect size of 0.5 to treat pain disease. Using this parameter from G*Power 3.1, with an 80% statistical power, alpha of 0.05, measuring six measures of three intervention groups. Therefore a sample size of 15 subjects with muscular TMD will be utilized. Subjects are from database of Occlusion and TMJ Center of Dentistry Faculty of Federal University of Bahia.

Randomization The subjects will be allocated consecutively to randomization as intervention order using the tool from randomization.com website (Dallal GE, http://www.randomization.com). The investigators will use the second generation suggested for crossover studies.

6.2 Materials The materials are available on the budget table and the questionnaire is annexed.

6.3 Data Collection Procedure All subjects will be treated using three different interventions (groups I1, I2 e I3) respecting the washout period of 7 days to avoid residual effects. The intervention order will be determined by randomization per group of intervention.

After COAT institutional authorization, subjects will be contact by phone and asked if they want to participate in the study. Those who wish to participate and qualify according to the selection criteria after completing the pre-screening questionnaire will be scheduled after reading and signing the consent form (2 copies). Women of chill-bearing potential will be required to take a urine pregnancy test during screening process. If a subject becomes pregnant during the course of the study, she will be withdrawn from the study. At the end of the first appointment the subject will take a VAS and ISTA diary home to complete 7 days before the baseline evaluation. The investigators will use the average of VAS and ISTA diary to get the baseline values.

During the second visit, all clinical and neurological assessments will be performed before and after tDCS stimulation. During the second visit (T2) clinical and neurological assessments will be performed. The clinical assessments will be guided by RDC/TMD, pain and anxiety diary and by sensory tests (Von Frey monofilaments and algometry/EMG system). The neurophysiological assessment will be done using EEG to analyze cortical activity. Each patient will be clinically and neurologically assessed before and after the stimulation, allowing data to be collected 6 times (T2 to T7) and also at the first visit.

To group I1, the parameters used in the TDCS will be 1mA with cathodal over the right DLPFC and anodal stimulation in the supraorbital contralateral area. With this chosen area the investigators aim to reach cerebral regions responsible for anxiety. To group I2, the same parameters will be used; however the current will be 2mA. The parameters to group I3, which is the control group, will be the same as the active and the device in sham mode. To acquire a placebo effect, the current will be used for the first 30 seconds and then reduced gradually until zero in 20 seconds. This method has been shown effective in previous studies and accepted by the academic community to blind subjects without any type of effects in the cortical excitability.

The current will be applied using 35cm2 electrodes soaked in saline substance (140mMol de NaCl water dissolved Mille-Q). The electrodes will be connected in the device driven by a 9v batteries and will be regulated by a digital multimeter (EZA EZ 984, China) standard error of ±1.5% (Montenegro et al., 2012).

All subjects will receive just one stimulation session for each type of intervention (I1, I2, I3), totaling 3 sessions. After tDCS sessions the subject will answer an adverse effects questionnaire. A trained researcher will do each procedure. A researcher responsible for the general coordination (E.P.S.) will hold the randomization list and just the responsible for the tDCS stimulation would know this information.

6.4 Study Variables Dependent: Visual Analogic Scale to pain, inventory of state-trit anxiety, sensory testing, TMS and EEG.

Independent: Cathodal tDCS over DLPFC (1mA/2mA) and placebo treatment. 6.5 Data Analysis Data will be recorded at an Excel 2010 sheet to be analyzed by a biostatistics professional who will not have access to randomization process. To verify improvements after tDCS session from each intervention group the investigators will use correlation test, post-hoc (to multiples compare), a parametric one-way ANOVA if the data distributions are normal or non-parametric if not normal and an intraclass concordance test. The difference among groups will be analyzed by a multiple variance analysis (placebo vs. 1mA, Placebo vs. 2mA and 1mA vs. 2mA) and p-value will be corrected to multiple compare (Bonferroni) to acquire a 0.05 significance level. All data will be analyzed by intention to treat.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-60 years, both male and female
* Having a diagnosis of muscular pain DTM according to IA and IB, axis I RDC/TMD
* Visual analogic scale (VAS) score from 4 to 10 for six months or longer
* Inventory of state-trit anxiety (ISTA) score more than 42

Exclusion Criteria:

* Pregnancy;
* Contraindications to tDCS:

  * metal implants
  * implanted brain devices
* History of alcohol or drugs abuse within the past 6 months as self-reported
* Use of carbamazepine within the past 6 months as self reported
* Any history of epilepsy, stroke, moderate-to-severe traumatic brain injury or severe migraines
* History of neurosurgery as self-reported
* History of joint problems as disc displacement, arthralgia, osteoarthritis and osteoarthritis (Axis I, II and III diagnosis)
* History of major psychiatric disorders such as schizophrenia and bipolar disorder
* Any other previously diagnosed disorder with symptoms similar to the DTM, such as fibromyalgia.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2014-07; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Visual Analogic Scale | 4 weeks
  The visual analogic scale allows us to convert subjective sensations as pain on numerical data. A 10cm scale where 0cm is no pain and 10cm the worse imaginable pain, will be used and the subjects will be asked to mark a point on the scale representing their pain. This instrument will be used by the subjects everyday during one week in a pain diary. A weekly response average will be calculated before the first interventions and after each one. Subjects will also fill a VAS before and after each tDCS session. The averages will be used to compare the VAS values before and after each intervention.

SECONDARY OUTCOMES:
Change from baseline in Electroencephalogram (EEG) | 4 weeks
  Another type of assessment is the electroencephalography, which measures the brain electrical current intensity using the analysis of waves. The alpha wave is related with relaxation and it is higher when the subject keeps her/his eyes closed, and lower when the eyes are open. The same can be seen in relaxation and alert states respectively. The EEG is a powerful tool to assess changes related to anxiety. The increase of alpha indicates reduction of chronic jitters (Hammond (2005).
  In this study a 24 channels EEG will be used associated with TMS, both according the international system 10x20 of electrodes. We will check alpha amplitudes before and after tDCS stimulation to see if the alpha waves will increase/decrease. The reference electrodes will be placed in the left ear lobe and in the masseter assessed spot. The data will be analyzed by MATLAB (The Mathworks, Inc., Natick, Massachusetts, USA) after the signals had been filtered from 0.1 to 35Hz and digitalized in 1450Hz.

OTHER OUTCOMES:
Pressure-pain threshold (PPT) | 4 weeks
  Pressure-pain threshold (PPT): PPT will be determined using blunt pressure delivered by a 1-cm2 hard-rubber probe using an approved device (EMG system). During testing, a series of discrete pressures are applied to the more painful masseter tender point (right or left side) with the control site being the right or left thenar area (non-painful site). The patient will let the investigator know when he/she feels any pain and at that time, the procedure will be stopped and the value will be recorded. This procedure will be repeated 3 times. The test will take approximately 7-10 min to complete. To use the same tender point we will make a template over masseter area.
Mechanical perception and pain threshold | 4 weeks
  Mechanical perception and pain threshold: will be tested on the thenar area using Semmes-Weinstein monofilaments (0,008 a 300g/mm2). Monofilament applications will be at the same points as the PPT assessments. The hairs will be applied until subject perceives the stimulus (sensory perception threshold) and describes it as painful (pain threshold). The threshold will be taken as the lowest force that causes sensory/pain perception
Inventory of State-Trait Anxiety | 4 weeks
  Inventory of State-Trait Anxiety (ISTA) The inventory of state-trit anxiety is used to evaluate objectively both aspects of anxiety, trait and state. When analyzing the trait we sought to evaluate the personality, auto image, the way one view a non-threatening situation as a true threat (Is that what you are trying to say?). State anxiety is the transitory emotional state, in response to environmental stimuli such as tachycardia, sweating, nausea and cramps. The questionnaire addresses 20 possible sensations. 40 answers we can acquire values from 1 to 4, where 1 is never, 2 sometimes, 3 often e 4 always. At the end the sum of all the answers will direct us to the scale results which are: normality (38-42), depression (>42) or anxiety (<38).

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo P Sena, PhD, Study Director — Federal University of Bahia; Rivail A Brandao, Master, Principal Investigator — Federal University of Bahia
Locations (1):
- Federal University of Bahia, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: Yes
We will send a report to each subject

REFERENCES:
- [Derived] Brandao Filho RA, Baptista AF, Brandao Rde A, Meneses FM, Okeson J, de Sena EP. Analgesic effect of cathodal transcranial current stimulation over right dorsolateral prefrontal cortex in subjects with muscular temporomandibular disorders: study protocol for a randomized controlled trial. Trials. 2015 Sep 17;16:415. doi: 10.1186/s13063-015-0938-0. PMID 26381733